CLINICAL TRIAL: NCT04737655
Title: Non-inferiority Evaluation of Trimbow in Critically Ill Patients Admitted in ICU Compared to Standard of Care
Acronym: TRIMICU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PARZIBUT Gilles (Other)
Responsible Party: Sponsor-Investigator, PARZIBUT Gilles, MD, adjoint head of clinics in university hospital of liege, departement ICU, University of Liege
Organization: University of Liege (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B7072020000051
Record Dates: First submitted 2021-01-07; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: COPD Exacerbation
MeSH Terms: interventions — Formoterol Fumarate; Glycopyrrolate

STUDY DESIGN:
Intervention Model Description: The study population will consist of one cohort of patients admitted in our hospital (CHU DE LIEGE) for acute exacerbation of COPD. The COPD has to be diagnosed based on the international recommendations (GOLD recommendations). The patient has to suffer from an acute severe exacerbation requiring an ICU stay of at least 24hours.
  Patients will be separated in 2 randomized groups (Trimbow + SOC versus SOC) 1:1.
  A total of 200 patients will be randomized in this study following the inclusion and exclusions criteria.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TRIMBOW + Standard of care (Active Comparator): 1. Inclusion
     * Maintenance therapy (LAMA or LABA) for COPD
     * Age >18
     * Admission for AE of COPD
     * Signed Inform consent (see protocol attached)
     * Admitted in ICU >24h and less than 72h
  2. Exclusion
     * No CI for studied medication
     * Not treated with studied medication for at least 3 months
     * Admitted in ICU for AE of COPD within the past 3 months
     * Intolerance to studied medication
     * Hospitalized since >6 days
     * ARDS condition (PAFI <200)
     * Admitted in ICU >72H
     * Patient with severe asthma
     * The use of high dose of ICS as baseline therapy
     * Right/left heart failure
     * Immunocompromized
     * Acute myocardial infaction
     * Left heart insufficiency (LVEF<35%)
     * Stroke <6 months prior to hospital admission
  Patients will be separated in 2 randomized groups (Trimbow + SOC versus SOC) 1:1.
  Interventions: Drug: TRIMBOW® pressurised inhalation solution: Beclometasone dipropionate / formoterol fumarate /glycopyrronium 87/5/9 µg per inhalation
- standard of care (No Intervention)

INTERVENTIONS:
Drug: TRIMBOW® pressurised inhalation solution: Beclometasone dipropionate / formoterol fumarate /glycopyrronium 87/5/9 µg per inhalation — Evaluate Trimbow associated with the standard of care in comparison with the standard of care alone.
  Arms: TRIMBOW + Standard of care

SUMMARY:
Objective: To evaluate non-inferiority of Trimbow, an approved therapy for treatment of severe COPD, in ICU compared to the standard of care which is based on the same therapeutic approach.

Study location: CHU Sart-Tilman, 4000 Liège, Belgium Study duration: 2 years

Type : Interventional

Methodology: Prospective clinical trial Number of patients: 200 (randomized 1:1)

Main Inclusion criteria :

* Maintenance therapy (LAMA or LABA) for COPD
* Age >18
* Admission for AE of COPD
* Signed Inform consent
* Admitted in ICU >24h

DETAILED DESCRIPTION:
In the ICU, the standard of care is still focused on the use of aerosolized therapies. These therapies are time consuming and largely used unless the lack of proven superiority in comparison with Pressurised metered dose inhalers (pMDIs) which are as effective and easier to use. Moreover, aerosolized therapies are associated with an increased risk of oropharyngeal deposition and not always efficiently delivered.

The use of new ventilation techniques like high flow canula oxygen therapy is also challenging in the particular context of inhaled therapies. Nowadays, no data are available to confirm the appropriate deposition of the inhaled therapies. Therefore, it's necessary to have to move forward the evaluation of pMDIs in the particular context of non invasive ventilation (for example with high-flow nasal oxygen therapy).

As the use of triple therapy is now the standard of care in COPD patients experiencing a severe exacerbation, it is the objective to propose the introduction of Trimbow as soon as possible following the onset of a severe exacerbation, even in critically ill patients.

3 Study objectives

3.1 Main objective

Evaluate the non inferiority of Trimbow associated with the standard of care in comparison with the standard of care alone.

3.2 Secondary objectives

Evaluate the other ICU-stay outcomes and long term outcomes of the patients.

4 Type of Study

An open label, prospective randomized trial

Phase A : Open label, prospective study in hospital. Shift in phase IV at hospital discharge (reimbursed treatment in Belgium, use of Trimbow as recommended)

Phase B : Trimbow prescribed as accepted in Belgium following reimbursement criteria : observational study (12 months), out of hospital. One visit in hospital every 3 months (as usual) with classical evaluation during the visit (clinical, functional, symptomatic, scales, exacerbation) 5 Study population

The study population will consist of one cohort of patients admitted in our hospital (CHU DE LIEGE) for acute exacerbation of COPD. The COPD has to be diagnosed based on the international recommendations (GOLD recommendations). The patient has to suffer from an acute severe exacerbation requiring an ICU stay of at least 24hours.

Patients will be separated in 2 randomized groups (Trimbow + SOC versus SOC) 1:1.

A total of 200 patients will be randomized in this study following the inclusion and exclusions criteria.

The study will be spited in 2 phases:

* Phase A: Hospitalization (interventional)
* Phase B: Follow up study after discharged (observational)

Investigational therapy TRIMBOW® pressurised inhalation solution: Beclometasone dipropionate / formoterol fumarate /glycopyrronium 87/5/9 µg per inhalation

Reference therapy DUOVENT®: Fenoterol 50 microg/ipratropium 20 microg (400/160 per day to 800/320 per day) Plus FLIXOTIDE®: fluticasone propionate (250-100 microg/day)

Administration Informed consent: our study falls within the context of the law governing clinical studies and requires the signature of an informed consent which will be duly signed with the presence of an investigator and after the patient or his legal representative has been able to ask the set of his questions.

Practical aspects At admission in our hospital, the patient or its legal representative will be asked to participate in the TRIMICU study. All the explanations will be given by the data manager in charge of the study. After a period of reflection, a local investigator will re-consider the different aspects of the study with the various stakeholders and will personally supervise the signing of the informed consent.

After signature, the patient will be randomized to trimbow + SOC versus SOC alone. Patients will be randomized in groups of 20 patients 10/10 by the study director or the data nurse. None of them will have any therapeutic contact with patients.

Once started, the patient will be followed daily by the data manager during his hospitalization (via study of the computerized file) and once every 3 months after his discharge from hospitalization by telephone contact and a follow-visit every 3 months.

Phase A:

Composite primary endpoint At ICU discharge: non inferiority of Trimbow + SOC versus SOC alone

* ICU Length of stay
* Time of Ventilation

At hospital discharge

- In hospital length of stay

Phase B Explore the survival rate without exacerbation at 1 year.

Safety variables Trimbow is known to be efficient in the specific case of severe COPD which is by definition the case of all COPD patients admitted in ICU. As it is the standard of care per se for ambulatory patients, treating patients earlier with this specific therapy designed for COPD patients is theoretically appropriate. Trimbow is compound of bronchodilators and inhaled corticosteroids already used in the specific ICU onset. No safety issue is expected for this specific study.

Safety variables

* Pneumonia
* Time of mechanical ventilation
* Need for invasive mechanical ventilation
* Ventilator-acquired pneumonia (VAP)
* Tachyarythmia
* Myocardial infarction

Statistical analysis Two primary endpoints were considered for the sample size determination: (1) the length of hospitalization stay (days) during Phase I, and (2) the survival rate (%) without exacerbation at 1 year during Phase II. It was found that a total of 200 patients (including a 15% drop-out rate) randomized in two groups of 100 subjects would be necessary to show the non-inferiority of the "SOC+Trimbow" treatment compared to "SOC alone" treatment with a power of 80% and an overall significance level of 5% for the two outcomes, by using two one-sided unpaired t-test at α=0.025. In the power calculation, a non-inferiority margin of 2 days was assumed for the hospitalization length of stay and of 5% for the survival without exacerbation at 1 year.

Statistical Methods Descriptive statistics will be performed for each continuous variable measured and will include mean, median, standard deviation, minimum, maximum and number of available observation. Frequency distributions will be used for ordinal and nominal variables and will include numbers and percentages of each of the scores or categories, and the number of missing observations.

All variables will be compared between control group (SOC alone) and test group (SOC + Trimbow) with the convenient statistical test. The primary outcomes i.e. survival without exacerbation at 1 year and length of hospitalization stay, will be compared with a non-inferiority test.

Statistics will be done on the maximum available data. Results will be considered significant at the 5% level (p<0.05). Calculations will be done with SAS version 9.4 and R.

Data anonymization and Security Each subject in the study will be assigned a unique subject number and will keep that number throughout the study. The medical investigators will keep a list linking the subject's number to the subject's names. He will follow all applicable privacy laws in order to protect a subject's privacy and confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance therapy (LAMA or LABA) for COPD
* Age >18
* Admission for AE of COPD
* Signed Inform consent (see protocol attached)
* Admitted in ICU >24h and less than 72h

Exclusion Criteria:

* No CI for studied medication
* Not treated with studied medication for at least 3 months
* Admitted in ICU for AE of COPD within the past 3 months
* Intolerance to studied medication
* Hospitalized since >6 days
* ARDS condition (PAFI <200)
* Admitted in ICU >72H
* Patient with severe asthma
* The use of high dose of ICS as baseline therapy
* Right/left heart failure
* Immunocompromized
* Acute myocardial infaction
* Left heart insufficiency (LVEF<35%)
* Stroke <6 months prior to hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the non inferiority of Trimbow associated with the standard of care in comparison with the standard of care alone. | 2 years
  Composite primary Endpoint associating the ICU Length of stay (in days) and Time of Ventilation (in days also)

SECONDARY OUTCOMES:
Assessment of the risk of exacerbation in the year. | 2 years
  number of exacerbations / year

IPD SHARING:
Plan to Share IPD: Undecided